CLINICAL TRIAL: NCT01105754
Title: A Multifaceted Prompting Intervention for Urban Children With Asthma
Acronym: PAIR-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jill Halterman, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25281; 1R01HL091835-01A1 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Parents of children in the standard care group will complete the baseline assessment, but no asthma prompt will be created for either the caregiver or provider, and no information regarding the interview will be shared with the provider. After the baseline assessment, the office visit will proceed according to usual care.
- Multifaceted Prompting Intervention (Experimental): Multifaceted Prompting Intervention
  Interventions: Behavioral: Multifaceted Prompting Intervention MPI

INTERVENTIONS:
Behavioral: Multifaceted Prompting Intervention MPI — Practices assigned to the MPI group will receive a simple prompt given to the provider at the time of the visit with information regarding the child's symptoms, medication use, environmental exposures, and recommendations for guideline-based preventive care. Practices will receive brief interactive seminars, resource guides, access to free asthma education programs, and practice-level feedback regarding their performance on key outcome measures.
  Caregivers will receive a simple prompt, community resources, and a blank asthma action plan form.
  Arms: Multifaceted Prompting Intervention

SUMMARY:
The overall goal of this project is to evaluate whether a multifaceted prompting intervention, administered in the urban primary care office setting, reduces morbidity among urban children with asthma. This study builds on our experience with a pilot study in two urban continuity clinics, in which we found that prompting clinicians about asthma severity and care guidelines at the time of an office visit resulted in improved preventive care delivery to inner-city children. This type of prompting program has the potential to substantially improve care for impoverished children with asthma, and we propose to establish: 1) whether these findings can be replicated in a similar study including a larger sample of urban children from different types of practices, and 2) whether the positive effects can be enhanced by more specific prompting directed towards both the provider and the caregiver and by providing practice-level supports and feedback. We hypothesize that children receiving a multifaceted prompting intervention (MPI) will experience less asthma-related morbidity (defined by symptom-free days at the 2-month follow-up) compared to children receiving usual care. Our secondary hypothesis is that children receiving the MPI will receive improved preventive asthma care (defined by guideline-based corrective actions taken at the index visit) compared to children receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* Mild persistent or more severe asthma severity, or poor asthma control
* Age >2 and <12 years.
* Parent or caregiver must give permission to the study, and children >7 will must provide assent.

Exclusion Criteria:

* Inability to speak and understand English or Spanish
* No access to a working phone for follow-up surveys
* The child having other significant medical conditions,
* Children in foster care or other situations in which consent cannot be obtained from a guardian.
* Prior enrollment in the study.
* Child will not be seen by a physician or nurse practitioner during their visit

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 638 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S. Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Fagnano M, Berkman E, Wiesenthal E, Butz A, Halterman JS. Depression among caregivers of children with asthma and its impact on communication with health care providers. Public Health. 2012 Dec;126(12):1051-7. doi: 10.1016/j.puhe.2012.08.007. Epub 2012 Oct 25. PMID 23102501
- [Background] Yee AB, Fagnano M, Halterman JS. Preventive asthma care delivery in the primary care office: missed opportunities for children with persistent asthma symptoms. Acad Pediatr. 2013 Mar-Apr;13(2):98-104. doi: 10.1016/j.acap.2012.10.009. Epub 2013 Jan 5. PMID 23294977
- [Background] Gutierrez SJ, Fagnano M, Wiesenthal E, Koehler AD, Halterman JS. Discrepancies between medical record data and parent reported use of preventive asthma medications. J Asthma. 2014 May;51(4):446-50. doi: 10.3109/02770903.2013.878351. Epub 2014 Jan 30. PMID 24404799
- [Background] Lewis P, Fagnano M, Koehler A, Halterman JS. Racial disparities at the point of care for urban children with persistent asthma. J Community Health. 2014 Aug;39(4):706-11. doi: 10.1007/s10900-013-9815-5. PMID 24435717
- [Background] Carlin C, Yee AB, Fagnano M, Halterman JS. The influence of Hispanic ethnicity on parent-provider communication about asthma. Clin Pediatr (Phila). 2014 Apr;53(4):380-6. doi: 10.1177/0009922813510598. Epub 2013 Nov 26. PMID 24281159
- [Result] Halterman JS, Fagnano M, Tremblay PJ, Fisher SG, Wang H, Rand C, Szilagyi P, Butz A. Prompting asthma intervention in Rochester-uniting parents and providers (PAIR-UP): a randomized trial. JAMA Pediatr. 2014 Oct;168(10):e141983. doi: 10.1001/jamapediatrics.2014.1983. Epub 2014 Oct 6. PMID 25288141
- [Derived] Goldstein NPN, Frey SM, Fagnano M, Okelo SO, Halterman JS. Identifying Which Urban Children With Asthma Benefit Most From Clinician Prompting: Subgroup Analyses From the Prompting Asthma Intervention in Rochester-Uniting Parents and Providers (PAIR-UP) Trial. Acad Pediatr. 2018 Apr;18(3):305-309. doi: 10.1016/j.acap.2017.08.015. Epub 2017 Sep 9. PMID 28899842

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Multifaceted Prompting Intervention
  Multifaceted Prompting Intervention MPI: Practices assigned to the MPI group will receive a simple prompt given to the provider at the time of the visit with information regarding the child's symptoms, medication use, environmental exposures, and recommendations for guideline-based preventive care. Practices will receive brief interactive seminars, resource guides, access to free asthma education programs, and practice-level feedback regarding their performance on key outcome measures.
  Caregivers will receive a simple prompt, community resources, and a blank asthma action plan form.
Period: Overall Study
Arm/Group | Standard Care | Intervention
Started | 319 | 319
Completed | 304 | 307
Not Completed | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Intervention | Total
Number analyzed (Participants) | 319 | 319 | 638
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.70 (2.9) | 6.72 (3.0) | 6.71 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 144 | 271
  Male | 192 | 175 | 367
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 126 | 103 | 229
  Not Hispanic or Latino | 193 | 216 | 409
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 103 | 127 | 230
  White | 77 | 74 | 151
  More than one race | 138 | 113 | 251
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 319 | 319 | 638

OUTCOME MEASURES:

1. Primary Outcome: Symptom Free Days
Description: The primary outcome is asthma morbidity measured by the number of symptom-free asthma days (SFD) reported over 2 weeks at the 2-month follow-up assessment.
Time Frame: 2 month follow-up assessment
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 297 | 300
Days | 9.5 (5.1) | 10.2 (4.8)

2. Secondary Outcome: Number of Children Who Received Guideline-based Asthma Care During the Intervention Visit.
Description: The number of children who received guideline-based asthma care (eg: inhaled steroid prescription, counseling for triggers, counseling for adherence) at the intervention visit based on parent interview at the 2-week follow-up and medical record review.
Time Frame: 2 week follow-up, and medical record review
Measure: Number; unit: participants
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 319 | 319
participants | 105 | 184

ADVERSE EVENTS:
Arm/Group | Standard Care | Intervention
Serious Adverse Events (participants affected / at risk) | 0/319 | 0/319
Other Adverse Events (participants affected / at risk) | 0/319 | 0/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No